CLINICAL TRIAL: NCT01943006
Title: Efficacy and Tolerability of Hirudoid Cream in Prophylaxis and Treatment of Superficial Infusion Thrombophlebitis
Brief Title: Efficacy and Tolerability of Hirudoid Cream in Prophylaxis and Treatment Infusion Phlebitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medinova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Hir-901113
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Thrombophlebitis; Phlebitis
Keywords: Mucopolysaccaride polysulfate (MPS); MPS; Heparinoide; Infusionphlebitis; Prevention; Superficial thrombophlebitis; Treatment
MeSH Terms: conditions — Thrombophlebitis; Phlebitis | interventions — mucopolysaccharide polysulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hirudoid cream (Experimental): Patient treated with Hirudoid cream 0.3% Mucopolysaccharide polysulfate
  Twice daily
  Interventions: Drug: Hirudoid cream 0.3 % Mucopolysaccharide polysulfate
- Placebo (Placebo Comparator): Patients treated with placebo cream without active substance
  Twice daily
  Interventions: Drug: Placebo cream without active substance

INTERVENTIONS:
Drug: Hirudoid cream 0.3 % Mucopolysaccharide polysulfate — Hirudoid cream
  Arms: Hirudoid cream
Drug: Placebo cream without active substance
  Arms: Placebo

SUMMARY:
Patients receiving nutritional emulsion for at least 3 days will be treated with Hirudoid cream or placebo cream to prevent and treat phlebitis caused by the infusion. The treatment is continued after the end of infusion for at least 7 days.

Number of patients developing superficial phlebitis and duration of phlebitis will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the hospital requiring to receive infusion of a complete nutritional emulsion for 3 days (Kabiven® Peripheral, 1400 kcal, 1920 ml, 750 mosmol/L, pH 5.6),
* Aged 18-65 years.
* Patients who are able to understand the requirements of the study and agree to sign an informed consent, approved by an Independent Ethic Committee (IEC)/Institutional Review Board (IRB), prior to the study.

Exclusion Criteria:

* Patients known to be allergic to Hirudoid or any ingredients of Hirudoid
* Patients with impaired skin integrity caused by lesion or soft tissue trauma
* Patients having skin lesions with ulcerations or any other severe dermatologic disease
* Patients has been received a complete nutritional emulsion infusion within 7 days of inclusion
* Patients with severe uncontrolled medical conditions, which makes it undesirable or unsafe for the patients to participate in the study, such as: Acute or chronic uncontrolled severe infections,Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction, serious uncontrolled cardiac arrhythmia or any other clinically serious cardiac disease, Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN; optimal glycaemic control should be achieved before starting trial therapy, Uncontrolled bleeding
* Patients known to have coagulation disorders such as Haemophilia, Thrombocytopenia, Thrombosis, Other severe hematologic conditions like leukaemia, especially with abnormal coagulation
* Patients who have symptoms of microangiopathy (small vessel disease) or neuropathy related to diabetes and other diseases
* Patients with hyperthyroidism and hypothyroidism
* Patients who are pregnant or breast feeding
* Patients who are on anticoagulant therapy (last 2 weeks)
* Patients with severe psychiatric conditions
* Patients who are unable to bear legal responsibility or unable to understand the study
* Patients who are unreliable or unable to comply with the protocol, like alcohol or drug abusers
* Patients who had been participated in another clinical trial in the past 12 weeks
* Patient is relatives of, or staff directly reporting to, the investigator
* Patient is employee of the sponsor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of patient developing superficial thrombophlebitis | 7 days

SECONDARY OUTCOMES:
Time to develop infusion related superficial thrombophlebitis | 7 days
Change of clinical symptoms in patients who developed superficial thrombophlebitis | 14 days
  Pain score (10-point visual analogue score) Extent of erythema
Time to complete resolution of signs and symptoms in patients who developed superficial thrombophlebitis | 14 days
Investigators' satisfaction | 14 days
  4-point rating scale
Patient' satisfaction | 14 days
  4-point rating scale
Number of adverse events | 14 days
  Number of any adverse events and adverse drug reactions including their severity experienced by the patients during the course of therapy
Global tolerability | 14 days
  Rating of tolerance by investigator and patients using targeted questionnaire 4-point scale (very good, good, moderate, no change or deterioration) at the end of the study

OTHER OUTCOMES:
Fasting blood glucose (FBS) | 14 days
  Laboratory test performed on day 1 and at the end of the study
Platelet, red blood cell and leukocyte count | 14 days
  Laboratory testing is performed on day 1 and end of study
Alanine transaminase (ALT), | 14 days
  Laboratory testing is performed on day 1 and end of study
Aspartate transaminase (AST), | 14 days
  Laboratory testing is performed on day 1 and end of study
Fibrinogen and activated partial thromboplastin time (aPTT) | 14 days
  Laboratory testing is performed on day 1 and end of study
Prothrombin time (PT) | 14 days
  Laboratory testing is performed on day 1 and end of study
Serum creatinine | 14 days
  Laboratory testing is performed on day 1 and end of study

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Siriraj Hospital, Bangkok
  - Chulalongkorn Hospital, Bangkok
  - Rajvithi Hospital, Bangkok
  - Bamrasnaradua Infectious Diseases Institute, Nonthaburi